CLINICAL TRIAL: NCT02864173
Title: Whole Genome Single Nucleotide Polymorphisms in Elderly Patients With Postoperative Cognitive Dysfunction
Acronym: GenPOCD
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Nicolai Goettel, MD, DESA, EDIC, University Hospital, Basel, Switzerland
Other Study IDs: GenPOCD
Record Dates: First submitted 2016-08-04; First posted 2016-08-11 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Postoperative cognitive dysfunction; Postoperative cognitive decline; Postoperative delirium; Cognitive outcome; Neuropsychology; Genetics
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood sample
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: Whole genome small nucleotide polymorphism genotyping

SUMMARY:
Postoperative cognitive dysfunction (POCD) presents as a long-lasting decline in cognitive function following surgery. Recognized as an important neuropsychological complication of anesthesia and surgery, POCD occurs predominantly in elderly patients, and even after minor procedures. It affects 41% of patients over the age of 60 years one week after major noncardiac surgery, and persists until the third postoperative month in 13% of cases. POCD has an adverse impact on quality of life, may result in prolonged hospitalization and increased health care costs, and is associated with the risk of leaving the labor market prematurely and dependency on social transfer payments, as well as increased one-year mortality. Elderly patients are particularly at risk. Other risk factors include a pre-existing cognitive impairment, cerebral, cardiac or vascular disease, diabetes, alcohol consumption and a lower level of education. The occurrence of postoperative delirium seems to predispose patients to POCD. However, POCD itself is not associated with the development of dementia.

The pathogenic mechanism leading to POCD remains unclear. Numerous etiologic pathways have been suggested: cerebral ischemia due to impaired intraoperative cerebral perfusion and/or oxygenation, systemic inflammation and the effect of proinflammatory cytokines on the brain, altered cholinergic neurotransmission, anesthetic neurotoxicity, hormonal changes induced by surgical stress, sleep or circadian disturbances, or genetic factors.

Several studies have explored possible associations between a specific genotype and POCD; however, these were predominantly performed in patients undergoing cardiac surgery or carotid endarterectomy. Previous reports primarily focused on the analysis of the apolipoprotein E genotype as a predisposing factor for POCD. Results of some of these studies have been pooled in a recent meta-analysis. Other studies have investigated polymorphisms of the human circadian clock gene HPER3, complement, cytochrome P450, platelet glycoprotein IIIa, phosphodiesterase 4D, P-selectin, C-reactive protein, and the inducible nitric oxide synthase promoter.

The primary aim of this retrospective study of available cohort data is to investigate a specific genotype and to identify single nucleotide polymorphisms (SNPs) which may predispose elderly patients undergoing major noncardiac surgery to POCD.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-IV
* Major noncardiac surgery under general anesthesia
* Native German or French speakers

Exclusion Criteria:

* Cardiac surgery
* Neurosurgery
* Surgery within 12 months prior to inclusion
* History of intracranial or cerebrovascular pathology
* Preoperative Mini-Mental State Examination (MMSE) score <24
* Psychiatric disease and long-term psychopharmacological treatment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged ≥65 years undergoing major noncardiac surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Consortium to Establish a Registry for Alzheimer's Disease Neuropsychological Assessment Battery (CERAD-NAB) scores at one week | Postoperative day 7

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) | Postoperative day 7
Trail Making Test Part A | Postoperative day 7
Trail Making Test Part B | Postoperative day 7
Phonemic Fluency Test (S-words) | Postoperative day 7

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Goettel, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No